CLINICAL TRIAL: NCT02785978
Title: Pilot Study to Evaluate ActiMyo Measured Activity in Parkinson Disease Patients & Healthy Volunteers
Acronym: Pre-QuantiPark
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut de Myologie, France (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Pre-QuantiPark
Record Dates: First submitted 2016-05-11; First posted 2016-05-30 (Estimated); Last update posted 2017-10-10 (Actual); Status verified 2017-10

CONDITIONS: Parkinson Disease; Healthy Volunteers
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Parkinson Disease Patients Group #1 (Experimental): PD patients with programmed levodopa challenge
  Interventions: Drug: Levodopa acute challenge; Other: Controlled environment tests (series of tasks of everyday life); Other: Standardized scales: MDS-UPDRS (Part II to IV) and RDRS; Device: ActiMyo recording; Other: Diary completion
- Parkinson Disease Patients Group #2 (Experimental): PD patients without programmed levodopa challenge
  Interventions: Other: Controlled environment tests (series of tasks of everyday life); Other: Standardized scales: MDS-UPDRS (Part II to IV) and RDRS; Device: ActiMyo recording; Other: Diary completion
- Healthy volunteers (Experimental): Healthy volunteers
  Interventions: Other: Controlled environment tests (series of tasks of everyday life); Device: ActiMyo recording; Other: Diary completion

INTERVENTIONS:
Drug: Levodopa acute challenge — Inclusion visit (simultaneous video + ActiMyo recording):
  Levodopa acute challenge and 2 hours of recording and medical monitoring
  Arms: Parkinson Disease Patients Group #1
Other: Controlled environment tests (series of tasks of everyday life) — Inclusion visit (simultaneous video + ActiMyo recording):
  Controlled environment tests (series of tasks of everyday life)
Other: Standardized scales: MDS-UPDRS (Part II to IV) and RDRS — Inclusion visit (simultaneous video + ActiMyo recording):
  Standardized scales: MDS-UPDRS (Part II to IV) and RDRS
  Arms: Parkinson Disease Patients Group #1; Parkinson Disease Patients Group #2
Device: ActiMyo recording — Continuous activity recording with ActiMyo during the 2 weeks of study participation
Other: Diary completion — Daily patient logbook completion during the 2 weeks of study participation

SUMMARY:
Pre-QuantiPark is a pilot study to evaluate the reliability and responsiveness of ActiMyo measured activity in PD patients. The purpose of the study is to provide validation of the ActiMyo, an innovative home-recording device enabling use in clinical trials and as an innovative tool for PD patient care.

ELIGIBILITY:
Patients:

Inclusion criteria

* Clinical diagnosis of idiopathic PD (UKPDSBB criteria)
* On stable parkinsonian medication regimen including levodopa for at least 4 weeks
* Male of female aged ≥18 years old
* Experiencing motor fluctuations and dyskinesia
* MoCA (Montreal Cognitive Assessment) ≥ 26
* Willing to adhere and comply to the protocol requirements as evi-dence by written informed consent
* Capable and willing to accurately using Actimyo
* Capable and willing to complete diaries
* Unlimited broadband internet access at home
* Agrees to be filmed
* Affiliated to or a beneficiary of a social security scheme
* PD patients subgroup #1 only: levodopa acute test scheduled as part of usual care

Exclusion Criteria

* Undergone surgery for the treatment of PD
* Apomorphine or Levodopa Pump in place
* Deep brain stimulation or transcranial magnetic stimulation
* Drug-induced parkinsonism
* Vascular parkinsonism
* Parkinson plus syndromes (such as multiple system atrophy, pro-gressive supranuclear palsy, and corticobasal degeneration)
* Other neurodegenerative disorders
* Any other significant medical or psychiatric illness that could inter-fere with study evaluation
* For women: pregnancy or current breastfeeding
* Under legal protection

Healthy subjects:

Inclusion criteria

* Male of female matched by age with PD patients ; aged ≥ 18
* Willing to adhere and comply to the protocol requirements as evi-dence by written informed consent
* Capable and willing to accurately using Actimyo
* Capable and willing to complete diaries
* MoCA (Montreal Cognitive Assessment) ≥ 26
* Unlimited broadband internet access at home
* Agrees to be filmed
* Affiliated to or a beneficiary of a social security scheme

Exclusion Criteria

* Any significant medical or psychiatric illness that could interfere with study evaluation
* For women: pregnancy or current breastfeeding
* Under legal protection
* Close or near relation of investigators, Institute of Myology employ-ees, or AFM-Telethon members.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Tremors measurement by ActiMyo® | Baseline
  PD patients only;
  1 to 3 hours of simultaneous video + ActiMyo® sensors recording and physician evaluation (tasks of every day life, MDS-UPDRS, RDRS and physician worksheet); Small steps will be detected and quantified following ActiMyo® raw data analysis and results will be compared to physician evaluation.
Small steps measurement by ActiMyo® | Baseline
  PD patients only;
  1 to 3 hours of simultaneous video + ActiMyo® sensors recording and physician evaluation (tasks of every day life, MDS-UPDRS, RDRS and physician worksheet); Small steps will be detected and quantified following ActiMyo® raw data analysis and results will be compared to physician evaluation.
Dyskinesia measurement by ActiMyo® | Baseline
  PD patients only;
  1 to 3 hours of simultaneous video + ActiMyo® sensors recording and physician evaluation (tasks of every day life, MDS-UPDRS, RDRS and physician worksheet); Dyskinesia will be detected and quantified following ActiMyo® raw data analysis and results will be compared to physician evaluation.

SECONDARY OUTCOMES:
Continuous home activity measurement by ActiMyo® | 2 weeks
  Subjects (PD patients and healthy volunteers) will wear ActiMyo® sensors everyday during 2 weeks and complete a hand-written paper diary to record their activity.
  Activity variables will be deduced from ActiMyo® raw data analysis.
Off, On without dyskinesia, on with dyskinesia states measurement by ActiMyo® | 2 weeks
  PD patients will wear ActiMyo® sensors everyday during 2 weeks and complete a hand-written paper diary to record their state (Off, On without dyskinesia, on with dyskinesia).
  Off, On without dyskinesia, on with dyskinesia states will be measured following ActiMyo® raw data analysis and compared to hand-written paper diary indicating states.
Everyday life tasks measurement by ActiMyo® | Baseline
  PD patients and healthy volunteers Every day life tasks will be measured following ActiMyo® raw data analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Teresa Gidaro, MD, PhD, Principal Investigator — Association Institut de Myologie
Locations (3):
- France (3):
  - Service de Neurochirurgie, Hopital Henri Mondor, Créteil
  - Association Institut de Myologie, Paris
  - Département des Maladies du Système Nerveux, GH Pitie Salpatriere, Paris